CLINICAL TRIAL: NCT05173233
Title: Confirmatory Clinical Study of Treating Tricuspid Regurgitation With K-Clip TM Transcatheter Annuloplasty System
Acronym: TriStar
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Huihe Medical Technology Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HH2021003
Record Dates: First submitted 2021-12-27; First posted 2021-12-29 (Actual); Last update posted 2022-04-21 (Actual); Status verified 2022-04

CONDITIONS: Tricuspid Regurgitation
MeSH Terms: conditions — Tricuspid Valve Insufficiency

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- K-clipTM transcatheter annuloplasty system (Experimental)
  Interventions: Device: Transcatheter Annuloplasty

INTERVENTIONS:
Device: Transcatheter Annuloplasty — Under echocardiography guidance, the transcatheter tricuspid annuloplasty system precisely reaches the specified position in the tricuspid valve region via jugular vein and superior vena cava approach. The enlarged tricuspid annular tissue is clamped with the clamp cpart and anchor part to reduce the perimeter of tricuspid annulus, so that the area of tricuspid orifice that could not be coapted is reduced. It plays the purpose of minimally invasive treatment of tricuspid valve.

SUMMARY:
The present clinical trial is performed to evaluate the effectiveness and safety of transcatheter tricuspid annuloplasty system manufactured by Shanghai Huihe Healthcare technology Co.,Ltd. for the treatment of subjects with severe or worse tricuspid regurgitation.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥60, male or female;
2. patients with severe or above secondary tricuspid regurgitation (TR≥4+) (secondary tricuspid regurgitation: tricuspid regurgitation caused by right atrial lesions, right ventricular cardiomyopathy, right ventricular myocardial infarction, left ventricular valvular disease, congenital heart disease and other diseases);
3. A multidisciplinary cardiac team (at least 2 doctors) consisting of cardiovascular physicians, cardiovascular surgeons, radiologists, anesthesiologists, etc., considered the subject to be at high risk for surgery and expected to benefit from tricuspid valve repair;
4. Left ventricular ejection fraction LVEF≥40%;
5. The subject voluntarily participates in the clinical trial and agrees or his/her guardian agrees to sign the informed consent.
6. Tricuspid regurgitation symptoms, such as chest tightness, asthma, shortness of breath, lower limb edema, ascites;
7. NYHA grade 2 to 4;
8. Patients who received tricuspid valve optimal drug therapy for ≥ 30 days were in stable condition;
9. In the case of the following diseases: mitral regurgitation, atrial fibrillation, coronary disease and heart failure, drug treatment should be ≥ 30 days or ≥ 30 days after instrumental treatment and the patient's condition is stable.

Exclusion Criteria:

1. patients with primary tricuspid regurgitation;
2. Patients with systolic pulmonary artery pressure ≥55 mmHg;
3. Patients with tricuspid valve or annuloplasty or tricuspid related procedure;
4. Patients with posterior tricuspid annulus calcification;
5. Evidence of mass, thrombosis or vegetations in the heart, jugular vein and superior vena cava;
6. patients with moderate or higher aortic stenosis, mitral stenosis, aortic regurgitation or mitral regurgitation;
7. patients with severely uncontrolled hypertension (systolic blood pressure ≥180 mmHg and/or diastolic blood pressure ≥110 mmHg);
8. Percutaneous coronary intervention within 1 month;
9. myocardial infarction or known unstable angina within 1 month;
10. Cerebrovascular accident within the past 3 months;
11. patients with active endocarditis or active rheumatic heart disease;
12. Patients with coagulation dysfunction, hypercoagulability or anemia (hemoglobin < 90 g/L);
13. patients with acute infection or other severe infection;
14. Patients with active peptic ulcer or active gastrointestinal bleeding;
15. severe end-stage diseases (such as malignant tumor, severe lung disease, liver disease, renal failure) with a life expectancy of less than one year;
16. Patients with known allergies or contraindications to the raw materials or drugs (such as antiplatelet drugs and anticoagulants) of the test products;
17. Persons addicted to alcohol, drugs or drugs;
18. Patients with cognitive impairment;
19. patients with histories of epilepsy or mental illness;
20. Participate in any other clinical trial (other than a registry study) within 30 days prior to signing the informed consent;
21. have a previous implantation of a pacemaker or defibrillator, or plan to implant a pacemaker or defibrillator;
22. Tricuspid stenosis;
23. Ebstain syndrome;
24. The anatomy of tricuspid annulus could not be assessed by TEE and TTE;
25. Hemodynamic instability;
26. chronic dialysis patients;
27. women who are pregnant during pregnancy, breast-feeding or during the clinical study;
28. Other conditions that the investigator considers inappropriate for participation in the clinical trial.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Estimated)
Dates: Start 2022-05-15 (Estimated); Primary Completion 2023-05-15 (Estimated); Study Completion 2027-05-15 (Estimated)

PRIMARY OUTCOMES:
All-cause mortality | 1-year after operation
Change of Tricuspid Regurgitation Grade | 1-year after operation
  Change of Tricuspid Regurgitation Grade assessed by corelab than baseline

SECONDARY OUTCOMES:
The success rate of post operation 12 months | 2 years, 3years, 4 years, 5 years
Success rate of device implantation | intra-procedure
Change in echocardiographic parameters | 1 month, 6 months, 1 year, 2 years, 3years, 4 years, 5 years
  Change in echocardiographic parameters：Tricuspid annulus A-P diameter（mm）、 Tricuspid annulus perimeter（mm）、Tricuspid annulus area(cm2)、Vena contracta width（mm）、EROA(cm2)、Regurgitation volume(ml)、IVC(mm)。
Change of Tricuspid Regurgitation Grade | 1 month, 6 months, 1 year, 2 years, 3years, 4 years, 5 years
NYHA | 1 month, 6 months, 1 year, 2 years, 3years, 4 years, 5 years
6 minutes walk distance | 1 month, 6 months, 1 year, 2 years, 3years, 4 years, 5 years
Kansas City Cardiomyopathy Questionnaire (KCCQ) | 1 month, 6 months, 1 year, 2 years, 3years, 4 years, 5 years

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Xu H, Chen M, Wang Z, Huo J, Li J, He F, Husanova F, Li H, Zhou D, Zhang X, Liu X, Song G, Li J, Luo J, Guo Y, Mou Y, Yuan S, Tao T, Wu S, Teng P, Ni Y, Ma L, Pan X, Ge J, Lee AP, Li W. Mid-Term Outcomes of K-Clip Transcatheter Tricuspid Annuloplasty System in Patients With Severe Functional Tricuspid Regurgitation. JACC Cardiovasc Interv. 2024 Dec 9;17(23):2796-2807. doi: 10.1016/j.jcin.2024.10.007. PMID 39663060
- [Derived] Xu H, Li W, Lee AP, Wu S, Husanova F, Wu B, Mou Y, Gu Y, Chen M, Tao T, Zhang Y, Zheng J, Yang A, Yuan S, Wang Q, Ni Y, Ma L. 30-Day Outcomes of Transcatheter Tricuspid Annuloplasty With the K-Clip System: A Single-Center, Observational Study. JACC Adv. 2023 Oct 27;2(9):100671. doi: 10.1016/j.jacadv.2023.100671. eCollection 2023 Nov. PMID 38938712
- [Derived] Wollborn J, Schuler A, Sheu RD, Shook DC, Nyman CB. Real-Time Multiplanar Reconstruction Imaging Using 3-Dimensional Transesophageal Echocardiography in Structural Heart Interventions. J Cardiothorac Vasc Anesth. 2023 Apr;37(4):570-581. doi: 10.1053/j.jvca.2022.11.011. Epub 2022 Nov 13. PMID 36517335